CLINICAL TRIAL: NCT01384500
Title: The Ornge Comparison of Tracheal Occlusion Pressures to Ensure Safety (OCTOPUS) Trial
Brief Title: The Ornge Comparison of Tracheal Occlusion Pressures to Ensure Safety Trial
Acronym: OCTOPUS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Workforce issues precluding study completion.
Sponsor: Ornge Transport Medicine (Other)
Responsible Party: Principal Investigator, Dr. Russell D. MacDonald, Medical Director, Ornge Transport Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 098-2011
Record Dates: First submitted 2011-06-20; First posted 2011-06-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Injury of Trachea; Friction and Pressure Injuries; Barotrauma; Transfer/Transport Injury
MeSH Terms: conditions — Pressure Ulcer; Barotrauma | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline in tube cuff (Experimental): Use of sterile saline to inflate tracheal tube cuff
  Interventions: Other: Saline in tube cuff
- Air in tube cuff (No Intervention): No intervention (control) - patient cohort, using air to inflate tracheal tube cuff.

INTERVENTIONS:
Other: Saline in tube cuff — Use of sterile saline, instead of air, to inflate tracheal tube cuff. Tracheal tube cuffs to be inflated to 22-25 cm H2O.
  Other Names: Sterile saline to inflate tracheal tube cuff.
  Arms: Saline in tube cuff

SUMMARY:
Patients who are intubated (breathing tube in windpipe) are often transported by air ambulance. Changes in atmospheric pressure during flight may cause pressure increases in the air-filled cuff holding the tube in the windpipe. Studies show that more than half the patients had potentially harmful pressures in the cuff during flight. High pressures lead to complications, such as injury to the windpipe. To avoid injury, cuff pressures must be kept at a safe level. There are many ways to avoid unsafe cuff pressures. One is to inflate the cuff with sterile fluid instead of air. Fluids are not subject to changes in atmospheric pressure. Using fluid, instead of air, in the cuff causes less pressure increases and less windpipe injury. The use and safety profile of this during transport by air ambulance has not been studied. This study compares tracheal tube cuff pressures, filled with air or fluid, at routine flying altitudes during patient transports by air ambulance.

DETAILED DESCRIPTION:
Introduction Air medical services routinely transport patients who are intubated and mechanically ventilated. Transporting this patient population is safe but patients subject to changes in barometric pressure in flight. Aircraft used typically maintain a cabin pressures of 3000 to 7000 feet above sea level. This compares to commercial aircraft that maintain cabin pressures of 5000 to 8000 feet. A known volume of gas will expand as the ambient pressure decreases. If the gas cannot expand, pressure exerted by the gas in an enclosed space will increase. An aircraft cabin with an ambient pressure of 3000 to 7000 feet altitude results in a 9 to 23% decrease in ambient pressure compared to sea level. Tracheal tube cuffs are subject to changes in ambient pressure that occur in transport. Tracheal tube cuffs minimize the risk of tracheal mucosal injury, but high pressures occur. A recent series of intubated adult patients undergoing transfer by helicopter showed that 58% had initial pressures greater than 40 cm H2O . A subsequent study revealed pressures exceeding 40 cm H2O in two thirds of patients and 30 cm H2O in nearly three quarters. There is a risk because tracheal mucosa blood flow is compromised at 30 cm H2O, and ceases at lateral wall pressures of 50 cm H2O. These high pressures can result in complications ranging from sore throat to major complications such as tracheal ischemia and fistula formation. To avoid tracheal injury and related complications, tracheal tube cuff pressures should be maintained at less than 30 cm H2O.

Sterile saline to inflate the cuff can decrease risk because it is not compressible or subject to atmospheric pressure changes as much as gases. Saline causes less cuff pressure increase and tracheal morbidity in the operating room, avoids excessive pressure due to changes in altitude, and is safe in transport. However, the ability of saline to prevent increases in cuff pressure in air medical transport and the safety profile of this use have not been studied.

Objectives Compare the tracheal tube cuff pressures, filled with either air or sterile saline, at altitudes routinely encountered when intubated and mechanically ventilated adult patients undergoing air medical transport.

Methods Study design Conduct a prospective, randomized, blinded study of tracheal tube cuff pressures, filled with either air or sterile saline, on pressurized fixed wing and unpressurized rotor wing aircraft to determine impact of cuff content (air versus saline) and altitude on cuff pressure in flight.

Study setting and population Ontario is a large Canadian province with a mix of urban, suburban, rural, and remote areas. Ornge Transport Medicine is the publicly funded air medical transport system providing all air medical patient transfers in Ontario. Ornge carries out approximately 19,000 patient transports annually, of which approximately 1,000 are intubated.

This study will screen all consecutive intubated patients transported by pressurized fixed wing aircraft and unpressurized rotor wing aircraft. Patients will be screened beginning July 1, 2011 and ending when the requisite number of patients have been receuited on each aircraft type. Patients will be eligible if they are adult (actual or estimated age >18 years), undergoing interfacility patient transfer, intubated with a cuffed tracheal tube and mechanically ventilated prior to transport, transported by an Ornge's dedicated aircraft and flight paramedic crew, with a planned flight of >20 minutes (rotor wing) or >30 minutes (fixed wing). Patients are excluded if they do not meet all inclusion criteria or have any condition that requires a cabin altitude of <1000 feet to prevent barotrauma. For ineligible patients, paramedics will submit the completed screening tool and copy of the patient care report to the research coordinator. Investigators will retrospectively review dispatch records to identify intubated patients who were transported to determine the total patient population eligible for this study. Planned flight times of >20 minutes (rotor wing) and >30 minutes (fixed wing) were selected because review of records for flights of lesser duration would not typically have enough time at cruising altitude to stabilize cabin pressure, equilibrate tracheal tube cuff pressure, and complete the in-flight portion of this protocol.

Study protocol This study will be conducted with two patient cohorts: 1) fixed wing patient cohort in pressurized cabin, and 2) rotor wing patient cohort in unpressurized cabin. Each cohort will be randomized to a 'sterile saline' ('experimental') or an 'air' ('control') arm. The paramedics will use a study-specific medical directive approved by the Ornge Medical Advisory Committee. Prior to commencing the study, paramedics will review a self-directed learning module. One investigator will contact each paramedic to confirm completion of the module and answer any questions. Paramedics will be able to enroll patients after the investigator confirms completion of the materials.

Paramedics will screen potentially eligible patients prior to departing from the sending facility, and randomize eligible patients. Patients withdrawn due to considerations of patient safety will not have a complete set of outcome data, but will be reported and analyzed separately.

Flight crew routinely determine the cabin altitudes unless there is a medical need for a cabin pressure equial to 1000 feet or less.

Randomization Randomization will occur by dedicated aircraft, in blocks of ten, with a 1:1 ratio. Study packages will be prepared, numbered sequentially, and tracked by a single Research Coordinator. The coordinator will maintain a confidential log of each package's randomization allocation, aircraft assignment, current location, and use. The coordinator will also receive all completed study materials and study data received from flight and paramedics crews, and all dispatch records to ensure all eligible patients were identified and screened by the paramedic crews.

Fixed wing Patients transported by pressurized fixed wing aircraft will be randomized to tracheal tube cuff filled with air or sterile saline. The cabin will be pressurized and set to maintain a fixed cabin pressure determined by the flight crew. All dedicated fixed wing aircraft are the same make and model capable of maintaining a fixed cabin pressure set.

Rotor wing Patients transported by unpressurized rotor wing aircraft will be randomized to tracheal tube cuff filled with either air or sterile saline. The cabin pressure on rotor wing aircraft is equivalent to that of the ambient air pressure because the cabin is not pressurized.

If a randomized patient experiences an unexpected situation that requires a cabin pressurization of 1000 feet above sea level or less at any point in the flight (either prior to or after measurement of tracheal tube cuff pressure at cruising altitude), the paramedic may request the pilot to pressurize the cabin according to patient requirements. If any medical condition or aviation situation requires deviation from the study protocol, management of the medical condition or aviation situation shall take precedence, and the patient may be withdrawn from the study. If a patient is randomized but does not complete the study, the patient will be withdrawn from the study, and the reasons will be reported in the "paramedic #1 data collection sheet". The patient will not included in the analysis of changes in tracheal tube cuff pressure if all pressure measurements were not completed, but the reason(s) for study termination will be reported.

Paramedics will complete their patient care report in the usual manner and fax it, along with the two paramedic data collection sheets, to the dedicated fax line using the "rapid fax transmission" cover page. They will then return all original documentation to Ornge corporate headquarters in the usual manner. The pilots will forward the pilot data collection sheet to Ornge Air corporate headquarters in the usual manner. All records are shipped and stored using policies and procedures consistent with existing privacy legislation and regulations. The research coordinator will enter all study data elements in a study-specific, password-protected database stored on a secure computer server.

Outcome measures The primary outcome measure is the incidence of tracheal tube cuff pressure exceeding 30 cm H2O during the cruise portion of flight. This is approximately 10 minutes after the aircraft has taken off. The secondary endpoints include the incidence of tracheal tube cuff pressure exceeding 30 cm H2O on initial inflation of the cuff prior to departure from sending facility, the change in cuff pressure from ground to in flight at cruising altitude, the incidence of cuff leak or other tracheal tube malfunction, and incidence of adverse events related to tracheal tube cuffs, (including those related to use of sterile saline in cuffs) in the transport setting. All outcome measures will be obtained and assessed on day 1, namely during the time period during which the flight paramedics are providing care for the patient. No data will be available after transfer of care takes place at the receiving facility.

Sample size and power calculations Tracheal tube cuff pressures are typically inflated to a pressure ranging from 20 to 25 cm H2O, with tracheal mucosal injury occurring at cuff pressures exceeding 30 cm H2O. Based on estimate of anticipated true difference in the means of cuff pressures on land and in flight of 12 and estimate of standard deviations of cuff pressure distributions, we will need to study 60 experimental subjects and 60 control subjects to be able to reject the null hypothesis that the mean change in cuff pressure of the experimental and control groups are equal with probability (power) 0.9. The type I error probability associated with this test of this null hypothesis is 0.05.

Assuming a completion rate of 0.75, we estimate it will take 160 enrolled subjects (80 air, 80 saline) on each aircraft type to obtain the needed number of patients. Ornge transports approximately 1,000 intubated and mechanically ventilated patients each year, of which approximately 35% are transported by fixed and 65% by rotor wing. It take 4 to 6 months to complete the study in the fixed wing patient population, and 2 to 3 months in the rotor wing population.

Data analysis Tracheal tube cuff pressures will be analyzed and reported as continuous variables. The presence of tracheal tube cuff pressures exceeding 30 cm H2O is a dichotomous outcome and reported as a proportion of those exceeding this threshold. Differences in mean change in tracheal tube cuff pressures between study groups (air or saline) within each aircraft type (rotor or fixed wing) will be reported as mean + standard deviation, and compared using the unpaired t test, with p<0.05 considered as significant. The relationship and strength of association between tracheal tube cuff pressures and altitude will be analyzed by regression by least squares methods and Pearson's correlation coefficient, respectively. The incidence of adverse events due to tracheal tube cuffs, including those due to use of saline in cuffs, will be reported using descriptive statistics. Differences in adverse events between study groups (air or saline) within each aircraft type (rotor or fixed wing) will be compared using the unpaired t test. Results are reported as mean + standard deviation, with p<0.05 considered as significant.

The Data Safety Monitoring Board (DSMB) comprises three individuals intimately associated with air medical patient transport, with a research and statistical expertise to perform the interim analyses and monitor the study for patient safety and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* interfacilty patient transfer
* cuffed tracheal tube
* age equal to or greater than 18 years
* planned flight time >20 minutes (helicopter) / >30 minutes (fixed wing)

Exclusion Criteria:

* age less than 18 years
* other advaced airway (non-tracheal tube)
* scene response
* planned flight time less than 20 minutes (helicopter) / 30 minutes (fixed wing)
* medical condition that requires cabin altitude less than 1000 feet above ground level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the incidence of tracheal tube cuff pressure exceeding 30 cm H2O during the cruise portion of flight. | During cruise portion of flight, approximately 10-15 minutes after aircraft take-off.
  The flight paramedics will measure the tracheal tube cuff pressure during the cruise portion of flight, approximately 10-15 minutes after the aircraft has taken off.

SECONDARY OUTCOMES:
Incidence of tracheal tube cuff pressure exceeding 30 cm H2O on initial inflation of the cuff prior to departure from sending facility. | Prior to departure from sending facility
  The flight paramedics will measure the tracheal tube cuff pressure prior to departing the sending facility.
The change in cuff pressure from ground to in flight at cruising altitude. | During cruise portion of flight.
  The flight paramedics will measure the tracheal tube cuff pressure during the cruise portion of flight, approximately 10-15 minutes after the aircraft has taken off.
The incidence of cuff leak or other tracheal tube malfunction. | Any point during care
  The flight paramedics will identify if there has been a tracheal tube malfunction at any point during their care, from first patient contact at the sending facility, through the flight, and until transfer of care at the receiving facility.
Incidence of adverse events related to tracheal tube cuffs in the transport setting. | Any point during care.
  The flight paramedics will identify if there has been an adverse event related to tracheal tube cuff at any point during their care, from first patient contact at the sending facility, through the flight, and until transfer of care at the receiving facility.

CONTACTS AND LOCATIONS:
Overall Officials: Russell MacDonald, MD MPH, Principal Investigator — Ornge Transport Medicine
Locations (1):
- Ornge Transport Medicine, Mississauga, Ontario, Canada